CLINICAL TRIAL: NCT04339179
Title: INA-RESPOND Observational Research on Infectious Disease Outbreaks and Difficult Cases of Unidentified Etiology in Indonesia
Brief Title: Observational Research on Infectious Disease Outbreaks and Difficult Cases of Unidentified Etiology in Indonesia
Acronym: INA-ORCHID
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Responsible Party: Sponsor
Other Study IDs: INA107; U1111-1263-1317 (Other: WHO UTN Number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Infectious Disease
Keywords: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, sputum, urine, stool, nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will investigate suspected infectious diseases of unknown etiology prospectively during outbreaks and at healthcare facilities, and retrospectively through historical samples where no etiology was ever determined. The study is designed to rapidly, flexibly, and consistently respond to any potential scenario in Indonesia, and the data collected will provide needed insight into the landscape of infectious diseases in the country. By better understanding the infectious causes of outbreaks and difficult hospitalized cases, the Indonesian Ministry of Health will be able to more accurately and efficiently control infectious diseases and craft healthcare policies.

DETAILED DESCRIPTION:
This is a study to identify the causative agents and describe the clinical characteristics of infectious disease outbreaks and difficult cases of unidentified etiology in Indonesia. It is a retrospective and prospective observational study with an exploratory design. There will be no intervention to the participants that is intended to affect their SoC or clinical outcome.

Retrospective study activities will be ongoing throughout the duration of the study. The INA-RESPOND Reference Lab will perform research tests on various specimens collected as part of historical outbreaks and previous difficult cases where an etiology was never identified.

Prospective study activities will be initiated upon official request from health authorities and health facilities/institutions. Requests are expected to be filtered through and evaluated by the 19 active INA-RESPOND Network sites before inclusion in the study. Samples collected during outbreaks and from difficult cases of unknown etiology will be analyzed at the INA-RESPOND Reference Lab at their own pace. Results from any research tests will be shared with the requesting authorities as research-use-only and are not intended to alter standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult or child of any age hospitalized with a current episode of illness with a presumed infectious disease of unidentified etiology
2. Negative for Dengue virus infection by an antigen-based and antibody-based diagnostic test (i.e. NS1 antigen test and Dengue-specific IgM test)
3. Negative for Salmonella Typhi infection by Standard of Care testing (i.e. blood culture, Widal test, or Tubex rapid test)
4. Able to provide a documented informed consent
5. Agrees to the collection and storage of specimens for laboratory testing and/or future research (participants may decline storage of specimens for future research)
6. For Ongoing patients in outbreak situations: Referral from the MoH as part of a suspected or identified outbreak of infectious disease

Exclusion Criteria:

* Investigators' discretion for patient safety and well being

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult or child of any age, both men and women hospitalized with a current episode of illness with a presumed infectious disease of unidentified etiology or referral from the MoH as part of a suspected or identified outbreak of infectious disease from 19 active INA-RESPOND Network sites across Indonesia
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Karyana, MPH, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia
Locations (19):
- Indonesia (19):
  - Site 520: University of Udayana/Sanglah Hospital, Denpasar, Bali
  - Site 560: University of Diponegoro/ Dr. Kariadi Hospital, Semarang, Central of Java
  - Site 530: University of Indonesia/ Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta
  - Site 540: Penyakit Infeksi Sulianti Saroso Hospital, Jakarta, DKI Jakarta
  - Site 590: Persahabatan Hospital, Jakarta, DKI Jakarta
  - Site 660 RSUD Abdul Wahab Sjahranie, Samarinda, East Kalimantan
  - Site 700 - RSUD Dr.TC Hillers, Maumere, East Nusa Tenggara
  - Site 570: University of Airlangga/ Dr. Soetomo Hospital, Surabaya, East of Java
  - Site 600 : Adam Malik Hospital, Medan, North Sumatra
  - Site 650: Budi Kemuliaan Hospital, Batam, Riau Islands
  - Site 630: M. Ansari Saleh Hospital, Banjarmasin, South Kalimantan
  - Site 690 - RSUD Abepura, Jayapura, Special Region of Papua
  - Site 510: University of Padjajaran/ Dr. Hasan Sadikin Hospital, Bandung, West Java
  - Site 610 : RSU Kabupaten Tangerang, Tangerang, West Java
  - Site 680 - RSUD dr Soedarso, Pontianak, West Kalimantan
  - Site 670 - RSUD Dr. Zainoel Abidin, Banda Aceh
  - Site 640: St. Carolus Hospital, Jakarta
  - Site 550: University of Hassanudin/ Dr. Wahidin Sudirohusodo Hospital, Makassar
  - Site 580: University of Gadjah Mada/ Dr. Sardjito Hospital, Yogyakarta

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment period was from November 2020 through July 2022. The study was done at 2 hospitals in Indonesia.
Groups:
- Suspected COVID-19 Cases: Hospitalized participants with suspected COVID-19
Period: Overall Study
Arm/Group | Suspected COVID-19 Cases
Started | 185
Completed | 185
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Hospitalized participants with suspected COVID-19
Arm/Group | Suspected COVID-19 Cases
Number analyzed (Participants) | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 175
  >=65 years | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [33 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 185
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Indonesia | 185

OUTCOME MEASURES:

1. Primary Outcome: Confirm Etiologies Among Suspected COVID-19 Cases
Description: Hospitalized suspected COVID-19 participants were monitored for at least 7-14 days after enrollment. Laboratory tests such as blood culture, RDT Influenza, RDT Dengue, Tubex TF, serology, and molecular were done to identify the etiology.
Time Frame: at least 7-14 days after enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Suspected COVID-19 Cases
Number analyzed (Participants) | 185
Participants
  SARS CoV-2 | 151
  Other pathogens: | 21
  Unidentified pathogens | 13

ADVERSE EVENTS:
Time Frame: 48 hours after blood drawn or specimen collection up to 14 days
Description: Any untoward or unfavorable medical occurrence in a human subject that occurs within 48 hours of a study-related blood draw or specimen collection that is possibly, probably, or definitely related to the blood drawn or specimen collection. Any event outside of this 48 hours window period will not be considered an AE for this study.
  All death cases which were not related to the study-related blood draw or specimen collection will not reported either as AE nor SAE.
Arm/Group | Suspected COVID-19 Cases
All-Cause Mortality (participants affected / at risk) | 5/185
Serious Adverse Events (participants affected / at risk) | 0/185
Other Adverse Events (participants affected / at risk) | 0/185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT04339179/Prot_SAP_ICF_000.pdf